CLINICAL TRIAL: NCT05860166
Title: Development of a Scale and Psychometric Test for Evaluation of Neuromotor Development of Infants in the Neonatal Intensive Care Unit
Brief Title: Development of a Scale for Evaluation of Neuromotor Development of Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Nilay Comuk Balci, Pt, Phd, Assoc. Prof., Ondokuz Mayıs University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2022/117
Record Dates: First submitted 2023-04-26; First posted 2023-05-16 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Infant Development; Premature; Neurodevelopmental Disorders; Neonatal Disease; Motor Delay
MeSH Terms: conditions — Premature Birth; Neurodevelopmental Disorders; Infant, Newborn, Diseases; Psychomotor Disorders | interventions — Weights and Measures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- trial group (Experimental): The Clinical trial group consists of infants to whom the tests will be applied.
  Interventions: Other: Test Scale

INTERVENTIONS:
Other: Test Scale — Developing an Neurodevelopment Test for evaluating infants in their neonatal period.

SUMMARY:
Although the scales used so far provide information about the neuromotor progression of a single baby, it is thought that they are not sufficient to distinguish babies from each other, and it is thought that there is no assessment battery that will adapt to the knowledge in their conditions and the functional development of babies. Therefore, the aim of our study is to reveal the applicability and psychometric properties of the Neonatal Infant Motor Assessment Scale (NIMAS) test, which reveals the neurological and motor performance of infants hospitalized in the NICU, both as automatic responses and functional behavior.

DETAILED DESCRIPTION:
Evaluations in the neonatal period become extremely important in terms of early diagnosis, medical follow-up, and planning of necessary interventions. Considering the sensitive and unstable physiological conditions of term and preterm babies who need neonatal intensive care, the tests to be used in the evaluation should be of valid, reliable, and easily applicable standards. There are various neuromotor and neurobehavioral scales according to the purpose of use in the evaluation of the baby. These scales are used to detect disorders of the infant's central nervous system function, examine the relationship between neuromotor and behavioral functions, determine the risk of complications that may be encountered in the future, monitor the infant's development, and determine the effectiveness of the interventions. While rating scales focus on examining all aspects of behavioral performance, they provide a comprehensive assessment of higher neurological functions. These scales are used in the follow-up of premature babies receiving care in the neonatal intensive care unit and to determine the differences that may occur in their neurobehavioral development. It is stated that more specific neurological examinations are required for the diagnosis of neurodevelopmental problems that the premature baby may encounter in the long term or the evaluation of general movements (GMs) provides better predictive value. In addition, the fact that premature babies continue to mature by compensating for the deficiencies in the newborn period thanks to their high neuroplasticity ability makes it difficult to predict the neurobehavioral status of premature babies precisely. Although the scales used so far give information about the neuromotor progression of a single baby, it is thought that they are not sufficient to distinguish babies from each other. Today, it is thought that no evaluation battery will adapt to the knowledge of their conditions and the functional development of babies. Therefore, our study aims to reveal the applicability and psychometric properties of the Neonatal Infant Motor Assessment Scale (NIMAS) test, which reveals the neurological and motor performance of infants hospitalized in the NICU, both as automatic responses and functional behavior.

ELIGIBILITY:
Inclusion Criteria:

* Born between 24-42 weeks of gestational age,
* The baby's vital signs are stable on the day of the test.

Exclusion Criteria:

* To undergo surgery,
* to be in the early post-op period <7 days (the day of the tests),
* Receiving treatment for sepsis or intensive phototherapy,
* The baby is intubated and on a mechanical ventilator,
* Unstable vital signs and taking sedative drugs,
* Having a genetic syndrome,
* Having other medical conditions that may affect physiotherapy practice, such as multiple congenital anomalies, tracheoesophageal fistula, diaphragmatic hernia, congenital heart malformation, and/or necrotizing enterocolitis.

Ages: 1 Day to 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 68 (Actual)
Dates: Start 2022-03-16 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-25 (Actual)

PRIMARY OUTCOMES:
Neonatal Infant Motor Assessment Scale | through study completion, an average of 1 year
  To reveal the applicability of the Neonatal Infant Motor Assessment Scale (NIMAS) test, which reveals the neurological and motor performance of infants hospitalized in the NICU.

SECONDARY OUTCOMES:
Dubowitz Neurologocial Assessment | through study completion, an average of 1 year
  Neurodevelopmental Assessment of the infants in neonatal period.
Amiel-Tison Neurologocial Assessment | through study completion, an average of 1 year
  Neurodevelopmental Assessment of the infants in neonatal period.

CONTACTS AND LOCATIONS:
Overall Officials: Nilay Comuk Balci, Principal Investigator — Ondokuz Mayıs University
Locations (1):
- Nilay Çömük Balci, Samsun, Atakum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No